CLINICAL TRIAL: NCT07108309
Title: A Randomized, Open-label, Comparative Clinical Study of the Efficacy, Safety, Pharmacokinetics, and Immunogenicity of BCD-236 in Combination With Chemotherapy in Patients With Relapsed and/or Metastatic Triple Negative Breast Cancer
Brief Title: BCD-236 in Combination With Chemotherapy in Patients With Relapsed and/or Metastatic Triple Negative Breast Cancer
Acronym: AREAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCD-236-2
Record Dates: First submitted 2025-08-04; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-02

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-236 + Chemotherapy (CHT) (Experimental): Subjects will receive BCD-236 +CHT
  Duration of treatment: until disease progression or intolerable toxicity or EOS
  Interventions: Biological: BCD-236; Drug: Chemotherapy
- Chemotherapy (CHT) (Active Comparator): Subjects will receive CHT.
  Duration of treatment: until disease progression or intolerable toxicity or EOS
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Biological: BCD-236 — as an intravenous infusion
  Arms: BCD-236 + Chemotherapy (CHT)
Drug: Chemotherapy — CHT (at the investigator's discretion):

SUMMARY:
To study the efficacy, safety, pharmacokinetics and immunogenicity of BCD-236 in combination with chemotherapeutic agents (CHT) in 2nd and subsequent lines of therapy of subjects with relapsed and/or metastatic triple negative breast cancer (TNBC).

ELIGIBILITY:
Main Inclusion Criteria:

* Signed informed consent and the subject's ability to comply with the requirements of the Clinical Study Protocol.
* Age ≥18 years and <75 years at the time of signing the informed consent form.
* Histologically verified diagnosis (there are documented results of relevant studies) of TNBC: ER 0-2 points, PR 0-2 points or ER <1%, PR <1% (ASCO/CAP); HER2 (≤1+) or HER2 (2+) in the absence of amplification of the Her-2-neu gene by ISH.
* TNBC is progressive or relapsing on or after systemic therapy.
* The subject received at least 1 line of systemic therapy for locally advanced unresectable or metastatic TNBC, or she experienced a relapse / progressive disease during or within 6 months after completion of post-operative (adjuvant) chemotherapy.
* Confirmed AXL expression in tumor cells according to immunohistochemistry.
* Availability of fresh (obtained as part of screening or before its start, but after disease progression or relapse on the last line of therapy) and archival (obtained before disease progression or relapse on the last line of therapy, if available) tumor material samples suitable for immunohistochemical examination to determine AXL expression.
* Presence of at least 1 measurable tumor lesion according to RECIST 1.1. criteria for CIR.
* ECOG score 0-1.
* Life expectancy ≥ 4 months from the date of signing of the informed consent form in the opinion of the Investigator.

Main Exclusion Criteria:

* Indications for radical therapy or radiotherapy (excluding minor surgery or radiation therapy for palliative purposes).
* Active CNS metastases and/or carcinomatous meningitis. Subjects with brain metastases may participate in the study provided that the metastases have been adequately treated with surgery or radiotherapy, and if they have been clinically stable for at least 4 weeks prior to randomization (i.e. no neurological symptoms, no need for corticosteroids, and no lesions >1.5 cm) and no evidence of new or increasing CNS metastases. Patients with newly diagnosed CNS metastases during screening may not be included in the study.

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 24 weeks
  According to RECIST 1.1 criteria by the central independent review (CIR)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 51 and 102 weeks
  According to RECIST 1.1 criteria by the central independent review (CIR)
Overall survival (OS) | 102 weeks
Disease control rate (DCR) | 24 weeks
  According to RECIST 1.1 criteria by the central independent review (CIR)
Time to response | 24 weeks
  According to RECIST 1.1 criteria by the central independent review (CIR)
Duration of response | 24 weeks
  According to RECIST 1.1 criteria by the central independent review (CIR)

CONTACTS AND LOCATIONS:
Overall Officials: Arina V Zinkina-Orikhan, PhD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (47):
- Belarus (3):
  - Health Institution "Brest Regional Oncology Center", Brest
  - "Gomel Regional Clinical Oncology Dispensary", Homyel
  - Minsk City Oncology Center, Minsk
- Russia (44):
  - State Budgetary Institution of Healthcare of the Arkhangelsk Region "Arkhangelsk Clinical Oncology Dispensary", Arkhangelsk
  - Regional State Budgetary Healthcare Institution "Altai Regional Oncology Dispensary", Barnaul
  - SBHI "Chelyabinsk regional clinical center Oncology and nuclear medicines", Chelyabinsk
  - Budgetary healthcare institution of the Udmurt Republic "Republican clinical oncology dispensary named after Sergei Grigorievich Primushko of the Ministry of Health of the Udmurt Republic, Izhevsk
  - SBHI of the Kaluga Region "Kaluga Regional Clinical Oncology Center", Kaluga
  - State Autonomous Institution of Health "Republican Clinical Oncological Dispensary of the Ministry of Health of the Republic of Tatarstan named after prof. M.Z.Sigal", Kazan'
  - SBHI "Clinical oncological Dispensary № 1" of the Ministry of Health of the Krasnodar Territory, Krasnodar
  - Branch of company "Hadassah Medical LCC", Moscow
  - Federal State Budgetary Scientific Institution "Russian Scientific Center of Surgery named after Academician B.V. Petrovsky", Moscow
  - FSAEI of Higher Education "First Moscow State Medical University named after I.M. Sechenov" of the Ministry of Health of the Russian Federation, Moscow
  - FSAEI of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), Moscow
  - FSAI "National Medical Research Center for Therapeutic and Rehabilitation Center" of the Ministry of Health of the Russian Federation, Moscow
  - FSBI "Lopukhin Federal Research and Clinical Center of Physical-Chemical Medicine of Federal Medical Biological Agency", Moscow
  - FSBI "National Medical Research Center of Oncology named after N. N. Blokhin" of the Ministry of Health of the Russian Federation, Moscow
  - Joint Stock Company "Medsi Group of Companies", Moscow
  - JSC "Modern medical technologies", Moscow
  - Limited Liability Company "Moscow Center for Rehabilitation Treatment", Moscow
  - SBHI of the City of Moscow "Moscow Clinical Scientific and Practical Center named after A.S. Loginov of the Moscow City Health Department", Moscow
  - State Budgetary Institution of Healthcare of the City of Moscow "City Clinical Hospital named after S.S. Yudin of the Moscow City Health Department, Moscow
  - State Budgetary Institution of Healthcare of the City of Moscow "Moscow City Oncology Hospital No. 62 of the Moscow City Healthcare Department", Moscow
  - SAHI of the Nizhny Novgorod region "Research Institute of Clinical Oncology "Nizhny Novgorod Regional Clinical Oncological Dispensary", Nizhny Novgorod
  - FBHI of the Novosibirsk Region "Novosibirsk Regional Clinical Oncological Dispensary", Novosibirsk
  - FSBI "National Medical Research Center for Radiology" of the Ministry of Health of the Russian Federation, Obninsk
  - FSBI "National Medical Research Center of Radiology" of the Ministry of Health of the Russian Federation Medical Radiological Research Center named after A.F. Tsyb, Obninsk
  - Budget Healthcare Institution of the Omsk region "Clinical Oncological Dispensary", Omsk
  - FSBI "National Medical Research Center of Oncology" of the Ministry of Health of the Russian Federation, Rostov-on-Don
  - State budgetary institution of the Ryazan region "Regional clinical oncology dispensary", Ryazan
  - FSBEI of Higher Education "North-Western State Medical University named after I. I. Mechnikov" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - FSBI "National medical research center of Oncology named after N.N. Petrov" Of Ministry of Health of the Russian Federation, Department of Breast Cancer Surgery, Saint Petersburg
  - FSBI "National medical research center of Oncology named after N.N. Petrov" Of Ministry of Health of the Russian Federation, Research Division of Innovative Techniques in Medical Oncology and Rehabilitation Medicine, Saint Petersburg
  - LLC "NRC Eco-Safety", Saint Petersburg
  - LLC "VitaMed", Saint Petersburg
  - Private healthcare institution "Clinical hospital "RZD-Medicine" of the city of St. Petersburg", Saint Petersburg
  - Private medical institution "Euromedservice", Saint Petersburg
  - SBHI "St. Petersburg Clinical Scientific and Practical Center for Specialized Types of Medical Care (Oncological) named after N.P. Napalkov", Saint Petersburg
  - SBHI of St. Petersburg "City Clinical Oncology Dispensary", Saint Petersburg
  - State Budgetary Healthcare Institution Leningrad Regional Clinical Hospital, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "National Research Mordovian State University named after N.P. Ogarev", Saransk
  - SBHI Arkhangelsk Region "Severodvinsk City Clinical Hospital No. 2 for Emergency Medicine", Severodvinsk
  - State Budgetary Healthcare Institution "Tambov Regional Oncology Clinical Dispensary", Tambov
  - SAHI Republican Clinical Oncology Dispensary of the Ministry of Health of the Republic of Bashkortostan, Ufa
  - SBHI "Volgograd Regional Clinical Oncological Dispensary", Volgograd
  - SBHI of the Yaroslavl region "Regional Clinical Oncological Hospital", Yaroslavl
  - SAHI of the Sverdlovsk region "Sverdlovsk Regional Oncological Center", Yekaterinburg